CLINICAL TRIAL: NCT01736059
Title: A Pilot Clinical Trial of the Feasibility and Safety of Intravitreal Autologous Adult Bone Marrow Stem Cells in Treating Eyes With Vision Loss From Retinopathy
Brief Title: Clinical Trial of Autologous Intravitreal Bone-marrow CD34+ Stem Cells for Retinopathy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 906595; BMSCRetPilot (Other: Other)
Record Dates: First submitted 2012-07-25; First posted 2012-11-29 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-exudative Age-related Macular Degeneration; Diabetic Retinopathy; Retina Vein Occlusion; Retinitis Pigmentosa; Hereditary Macular Degeneration
Keywords: Stem cells; intravitreal; bone marrow CD34+ cells; retinal disease; clinical trial; autologous
MeSH Terms: conditions — Diabetic Retinopathy; Retinitis Pigmentosa; Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem cell treated (Experimental)
  Interventions: Drug: CD34+ bone marrow stem cells intravitreal

INTERVENTIONS:
Drug: CD34+ bone marrow stem cells intravitreal

SUMMARY:
This pilot study is to determine whether it would be safe and feasible to inject CD34+ stem cells from bone marrow into the eye as treatment for patients who are irreversibly blind from various retinal conditions.

DETAILED DESCRIPTION:
In this pilot clinical trial, eyes with irreversible vision loss from retinal degenerative conditions (macular degeneration or retinitis pigmentosa) or retinal vascular disease (diabetic retinopathy or retinal vein occlusion) will be treated with intravitreal injection of autologous CD34+ stem cells isolated from bone marrow aspirate under Good Manufacturing Practice conditions. This study will determine whether there are any major safety and feasibility concerns using this therapy. Patients will be followed for 6 months after treatment by serial comprehensive eye examination supplemented with various retinal imaging and diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years of age
* visual acuity 20/100 to CF
* duration of vision loss > 3 months
* vision loss from macular degeneration, retinitis pigmentosa, retinal vein occlusion or diabetic retinopathy
* the study eye has the worse visual acuity
* no active eye or systemic disease
* no history of macular edema or retinal/choroidal neovascularization requiring treatment within 6 months
* no significant media opacity
* no coagulopathy or other hematologic abnormality
* no concurrent immunosuppressive therapy
* able to keep follow-up for 6 months

Exclusion Criteria:

* allergy to fluorescein dye
* other concurrent retinal or optic nerve disease affecting vision

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-07; Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular adverse events | 1 day to 6 months
  As evident on eye examination by severe decrease in vision and/or adverse effect requiring major treatment intervention directly attributable to study treatment.

SECONDARY OUTCOMES:
The number of stem cells isolated and injected into the study eye | 1 day
  Will determine the yield of the bone marrow aspiration and stem cell isolation procedures.

OTHER OUTCOMES:
Incidence and severity of systemic adverse events | 1 day to 6 months
  Any systemic adverse event attributable to the bone marrow aspiration or intravitreal injection of the stem cells.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna s Park, MD PhD, Principal Investigator — University of California Davis Eye Center
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Once study is completed, the study findings will be published in peer reviewed publication for public access.

REFERENCES:
- [Background] Park SS. Cell Therapy Applications for Retinal Vascular Diseases: Diabetic Retinopathy and Retinal Vein Occlusion. Invest Ophthalmol Vis Sci. 2016 Apr 1;57(5):ORSFj1-ORSFj10. doi: 10.1167/iovs.15-17594. PMID 27116667
- [Result] Park SS, Bauer G, Abedi M, Pontow S, Panorgias A, Jonnal R, Zawadzki RJ, Werner JS, Nolta J. Intravitreal autologous bone marrow CD34+ cell therapy for ischemic and degenerative retinal disorders: preliminary phase 1 clinical trial findings. Invest Ophthalmol Vis Sci. 2014 Dec 9;56(1):81-9. doi: 10.1167/iovs.14-15415. PMID 25491299
- See also: Learn more or sign up for the study here! — https://studypages.com/s/innovative-stem-cell-study-for-serious-vision-loss-at-uc-davis-eye-center-906754/